CLINICAL TRIAL: NCT03990753
Title: Microbiome/Peptidome-based Model for Non-invasive Detection of High-risk Gastroesophageal Varices in Compensated Cirrhosis (CHESS1901/APPHA1901): A Prospective Multicenter Study
Brief Title: Microbiome/Peptidome-based Model for Non-invasive Detection of High-risk Gastroesophageal Varices in Compensated Cirrhosis (CHESS1901/APPHA1901)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Southern Medical University, China (Other); LanZhou University (Other); Zhongda Hospital (Other); Guangdong Second Provincial General Hospital (Other); Xingtai People's Hospital (Other); The Third Hospital of Zhenjiang Affiliated Jiangsu University (Unknown); Tianjin Second People's Hospital (Other); Zhejiang University Lishui Hospital (Unknown); The Second Hospital of Anhui Medical University (Other); The Sixth People's Hospital of Shenyang (Other); Xi'an Gaoxin Hospital (Other); King Chulalongkorn Memorial Hospital affiliated to Chulalongkorn University (Unknown); Ankara University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: CHESS1901
Record Dates: First submitted 2019-06-16; First posted 2019-06-19 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Compensated Cirrhosis
Keywords: Microbiome/Peptidome; High-risk Gastroesophageal Varices; Compensated Cirrhosis
MeSH Terms: interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall eligible participants: Eligible participants will receive standard esophagogastroduodenoscopy and microbiome/peptidome examination.
  Interventions: Diagnostic Test: esophagogastroduodenoscopy

INTERVENTIONS:
Diagnostic Test: esophagogastroduodenoscopy — standard esophagogastroduodenoscopy

SUMMARY:
Variceal hemorrhage is a lethal complication in patients with cirrhosis and portal hypertension. Identification of varices needing treatment in compensated cirrhosis is, therefore, of great therapeutic and prognostic importance. The gold standard for diagnosing gastroesophageal varices and evaluating the risk of variceal hemorrhage is esophagogastroduodenoscopy. According to the Baveno VI consensus, for those with high-risk varices (HRV), either non-selective beta blockers or endoscopic band ligation is recommended for the prevention of the first variceal bleeding. However, the invasiveness and uncomfortableness during the esophagogastroduodenoscopy procedure has hindered its use in clinical practice, especially in patients with compensated cirrhosis. Sufficient accurate non-invasive tools for detection of HRV are warranted to safely avoid the use of esophagogastroduodenoscopy.

Advanced technologies including next-generation sequencing and MALDI-TOF mass spectrometry have the potential to be applied in this field. The latter is a widespread adopted tool in clinical microbiology for rapid, accurate and cost-effective identification of cultured bacteria and fungi. Recently, microbiome and peptidome have been proved their roles in the end-stage liver disease (e.g. cirrhosis, hepatocellular carcinoma), which may exhibit predictive capacity of HRV. In the present study, the investigators aim to conduct a prospective, multicenter diagnostic trial in 12 sites in China, 1 site in Turkey and 1 site in Thailand to evaluate the diagnostic performance of the microbiome/peptidome-based model for HRV detection in compensated cirrhosis.

DETAILED DESCRIPTION:
Variceal hemorrhage is a lethal complication in patients with cirrhosis and portal hypertension. Identification of varices needing treatment in compensated cirrhosis is, therefore, of great therapeutic and prognostic importance. The gold standard for diagnosing gastroesophageal varices and evaluating the risk of variceal hemorrhage is esophagogastroduodenoscopy. According to the Baveno VI consensus, for those with high-risk varices (HRV), either non-selective beta blockers or endoscopic band ligation is recommended for the prevention of the first variceal bleeding. However, the invasiveness and uncomfortableness during the esophagogastroduodenoscopy procedure has hindered its use in clinical practice, especially in patients with compensated cirrhosis. Sufficient accurate non-invasive tools for detection of HRV are warranted to safely avoid the use of esophagogastroduodenoscopy.

Advanced technologies including next-generation sequencing and MALDI-TOF mass spectrometry have the potential to be applied in this field. The latter is a widespread adopted tool in clinical microbiology for rapid, accurate and cost-effective identification of cultured bacteria and fungi. Recently, microbiome and peptidome have been proved their roles in the end-stage liver disease (e.g. cirrhosis, hepatocellular carcinoma), which may exhibit predictive capacity of HRV. In the present study, the investigators aim to conduct a prospective, multicenter diagnostic trial in 12 sites (The First Hospital of Lanzhou University; Zhujiang Hospital of Southern Medical University; Nanfang Hospital of Southern Medical University; Xingtai People's Hospital; Zhongda Hospital, Medical School, Southeast University; The Third People's Hospital affiliated to Jiangsu University; Guangdong Second Provincial General Hospital; Tianjin Infectious Disease Hospital; Lishui Municipal Central Hospital; The Second Hospital of Anhui Medical University; Xi'an Gaoxin Hospital; The Sixth People's Hospital of Shenyang) in China, 1 site (Ankara University School of Medicine) in Turkey and 1 site (King Chulalongkorn Memorial Hospital affiliated to Chulalongkorn University) in Thailand to evaluate the diagnostic performance of the microbiome/peptidome-based model for HRV detection in compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years;
* confirmed compensated cirrhosis based on liver biopsy or clinical findings;
* without decompensated events (e.g. ascites, bleeding, or overt encephalopathy);
* scheduled to undergo esophagogastroduodenoscopy;
* estimated survival time> 24 months, and model for end-stage liver disease (MELD) score< 19, and without liver transplant;
* with written informed consent.

Exclusion Criteria:

* contradictions for esophagogastroduodenoscopy;
* use of antibiotics, prebiotics, probiotics and proton pump inhibitors within 3 months upon recruitment.
* pregnancy or unknown pregnancy status.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with compensated cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2022-06-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of microbiome/peptidome-based model for high-risk varices | 1 day
  Diagnostic performance of microbiome/peptidome-based model to determine the presence or absence of high-risk varices when compared with esophagogastroduodenoscopy as the reference standard

SECONDARY OUTCOMES:
Diagnostic performance of microbiome/peptidome-based model for decompensation or death | 3 years
  Diagnostic performance of microbiome/peptidome-based model to determine the presence or absence of decompensation (defined as development of ascites, bleeding, or overt encephalopathy) or death within 3-year follow-up
Diagnostic performance of microbiome/peptidome-based model for hepatic venous pressure gradient | 1 day
  Diagnostic performance of microbiome/peptidome-based model to determine the level of hepatic venous pressure gradient

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, PhD, Principal Investigator — Southern Medical University, China; Xiaolong Qi, MD, Principal Investigator — LanZhou University
Locations (14):
- China (12):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - Zhongda Hospital, Medical School, Southeast University, Nanjing, Jiangsu
  - The Third Hospital of Zhenjiang Affiliated Jiangsu University, Zhenjiang, Jiangsu
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - Xi'an Gaoxin Hospital, Xi’an, Shanxi
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - Zhejiang University Lishui Hospital, Lishui, Zhejiang
- King Chulalongkorn Memorial Hospital affiliated to Chulalongkorn University, Bangkok, Thailand
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] He Y, Wu W, Zheng HM, Li P, McDonald D, Sheng HF, Chen MX, Chen ZH, Ji GY, Zheng ZD, Mujagond P, Chen XJ, Rong ZH, Chen P, Lyu LY, Wang X, Wu CB, Yu N, Xu YJ, Yin J, Raes J, Knight R, Ma WJ, Zhou HW. Regional variation limits applications of healthy gut microbiome reference ranges and disease models. Nat Med. 2018 Oct;24(10):1532-1535. doi: 10.1038/s41591-018-0164-x. Epub 2018 Aug 27. PMID 30150716
- [Background] Qi X, Li Z, Huang J, Zhu Y, Liu H, Zhou F, Liu C, Xiao C, Dong J, Zhao Y, Xu M, Xing S, Xu W, Yang C. Virtual portal pressure gradient from anatomic CT angiography. Gut. 2015 Jun;64(6):1004-5. doi: 10.1136/gutjnl-2014-308543. Epub 2014 Nov 14. No abstract available. PMID 25398771
- [Background] Qi X, An W, Liu F, Qi R, Wang L, Liu Y, Liu C, Xiang Y, Hui J, Liu Z, Qi X, Liu C, Peng B, Ding H, Yang Y, He X, Hou J, Tian J, Li Z. Virtual Hepatic Venous Pressure Gradient with CT Angiography (CHESS 1601): A Prospective Multicenter Study for the Noninvasive Diagnosis of Portal Hypertension. Radiology. 2019 Feb;290(2):370-377. doi: 10.1148/radiol.2018180425. Epub 2018 Nov 20. PMID 30457484
- [Background] Liu F, Ning Z, Liu Y, Liu D, Tian J, Luo H, An W, Huang Y, Zou J, Liu C, Liu C, Wang L, Liu Z, Qi R, Zuo C, Zhang Q, Wang J, Zhao D, Duan Y, Peng B, Qi X, Zhang Y, Yang Y, Hou J, Dong J, Li Z, Ding H, Zhang Y, Qi X. Development and validation of a radiomics signature for clinically significant portal hypertension in cirrhosis (CHESS1701): a prospective multicenter study. EBioMedicine. 2018 Oct;36:151-158. doi: 10.1016/j.ebiom.2018.09.023. Epub 2018 Sep 27. PMID 30268833
- [Background] Wang FS, Fan JG, Zhang Z, Gao B, Wang HY. The global burden of liver disease: the major impact of China. Hepatology. 2014 Dec;60(6):2099-108. doi: 10.1002/hep.27406. Epub 2014 Oct 29. PMID 25164003
- [Background] Garcia-Lezana T, Raurell I, Bravo M, Torres-Arauz M, Salcedo MT, Santiago A, Schoenenberger A, Manichanh C, Genesca J, Martell M, Augustin S. Restoration of a healthy intestinal microbiota normalizes portal hypertension in a rat model of nonalcoholic steatohepatitis. Hepatology. 2018 Apr;67(4):1485-1498. doi: 10.1002/hep.29646. Epub 2018 Feb 19. PMID 29113028
- [Background] Hoyles L, Fernandez-Real JM, Federici M, Serino M, Abbott J, Charpentier J, Heymes C, Luque JL, Anthony E, Barton RH, Chilloux J, Myridakis A, Martinez-Gili L, Moreno-Navarrete JM, Benhamed F, Azalbert V, Blasco-Baque V, Puig J, Xifra G, Ricart W, Tomlinson C, Woodbridge M, Cardellini M, Davato F, Cardolini I, Porzio O, Gentileschi P, Lopez F, Foufelle F, Butcher SA, Holmes E, Nicholson JK, Postic C, Burcelin R, Dumas ME. Molecular phenomics and metagenomics of hepatic steatosis in non-diabetic obese women. Nat Med. 2018 Jul;24(7):1070-1080. doi: 10.1038/s41591-018-0061-3. Epub 2018 Jun 25. PMID 29942096
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365